CLINICAL TRIAL: NCT02933060
Title: Intravenous Fluid Therapy for the Treatment of Emergency Department Patients With Migraine Headache: a Pilot Randomized Controlled Trial
Brief Title: Intravenous Fluid Therapy for the Treatment of Emergency Department Patients With Migraine Headache
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The Cooper Health System (Other)
Responsible Party: Principal Investigator, Christopher Jones, Assistant Professor, The Cooper Health System
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16-133
Record Dates: First submitted 2016-10-12; First posted 2016-10-14 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Migraine Headache
Keywords: intravenous fluid; headache
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV fluid bolus (Experimental): Patients will receive a 1000 ml bolus of normal saline, administered over 60 minutes.
  Interventions: Other: Normal saline (1000 mL)
- Control (Sham Comparator): Patients will have an IV catheter and will be connected to an IV bag, but will receive only 10 ml of normal saline over 60 minutes.
  Interventions: Other: Control

INTERVENTIONS:
Other: Normal saline (1000 mL)
  Arms: IV fluid bolus
Other: Control
  Arms: Control

SUMMARY:
The purpose of this study is to determine whether patients in the emergency department with migraine headache who are administered an intravenous fluid bolus will report greater improvement in pain scores than control patients.

DETAILED DESCRIPTION:
The investigators intend to perform a small-scale pilot study assessing the effectiveness of IV fluid therapy for patients presenting to the ED with migraine headache. Patients will be randomly allocated to receive a bolus of 1000 ml normal saline or no fluid bolus. Patients and outcome assessors will be blinded to the assigned study group. Research assistants will assess pain scores, nausea, and functional disability at time 0 (just prior to starting the intervention), 60 minutes, and 120 minutes. Participants will be contacted 48 hours after leaving the ED to assess symptom burden following discharge.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Fluent in English
* Meets International Classification of Headache Disorders (3rd ed) criteria for migraine headache:

A. At least five attacks fulfilling criteria B-D B. Headache attacks lasting 4-72 hours (untreated or unsuccessfully treated)

C. Headache has at least two of the following four characteristics:

unilateral location pulsating quality moderate or severe pain intensity aggravation by or causing avoidance of routine physical activity (e.g. walking or climbing stairs)

D. During headache at least one of the following:

1. nausea and/or vomiting
2. photophobia and phonophobia E. Not better accounted for by another ICHD-3 diagnosis.

Exclusion Criteria:

* Intravenous Fluids are contraindicated in the opinion of the emergency department physician caring for the patient (ex patient has an exacerbation of congestive heart failure).
* Intravenous fluids are required in the opinion of the emergency department physician caring for the patient (ex patient has intractable vomiting, patient has severe dehydration).
* Have already received greater than or equal to 500 ml of intravenous fluid during this emergency department visit, prior to enrollment.
* Currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-01; Primary Completion 2017-09-26 (Actual); Study Completion 2017-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Jones, MD, Principal Investigator — Cooper Medical School of Rowan University
Locations (1):
- Cooper Univeristy Hospital, Camden, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jones CW, Remboski LB, Freeze B, Braz VA, Gaughan JP, McLean SA. Intravenous Fluid for the Treatment of Emergency Department Patients With Migraine Headache: A Randomized Controlled Trial. Ann Emerg Med. 2019 Feb;73(2):150-156. doi: 10.1016/j.annemergmed.2018.09.004. Epub 2018 Oct 26. PMID 30665504

RESULTS

PARTICIPANT FLOW:
Groups:
- IV Fluid Bolus: Patients will receive a 1000 ml bolus of normal saline, administered over 60 minutes.
  Normal saline (1000 mL)
- Control: Patients will have an IV catheter and will be connected to an IV bag, but will receive only 10 ml of normal saline over 60 minutes.
  Control
Period: Overall Study
Arm/Group | IV Fluid Bolus | Control
Started | 25 | 25
Completed | 25 | 24
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Fluid Bolus | Control | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 34 [25 to 40] | 37 [30 to 50] | 35 [28 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 22 | 41
  Male | 6 | 2 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 7 | 17
  Not Hispanic or Latino | 13 | 17 | 30
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 8 | 18
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 6 | 11
Baseline Verbal Pain Score; median (IQR) [Median (Inter-Quartile Range); unit: Units on a scale] — (0 = no pain, 10 = maximum pain)
  Units on a scale | 8 [7 to 10] | 9 [8 to 10] | 9 [7.5 to 10]

OUTCOME MEASURES:

1. Primary Outcome: Verbal Pain Score at 60 Minutes
Description: The primary outcome will be the difference in verbal pain rating (0 = no pain, 10 = maximum pain) between the start of the study intervention and one hour later, at completion of the intervention. The minimum clinically significant difference between treatment groups on the 0-10 verbal scale is 1.3.
Time Frame: 60 minutes
Measure: Mean (95% Confidence Interval); unit: units on a scale (0-10)
Arm/Group | IV Fluid Bolus | Control
Number analyzed (Participants) | 25 | 24
units on a scale (0-10) | 4.5 [3.7 to 5.3] | 4.9 [3.5 to 6.2]

2. Secondary Outcome: Verbal Pain Score at 120 Minutes
Description: The difference in verbal pain rating (0 = no pain, 10 = maximum pain) between the start of the study intervention and 2 hours later. The minimum clinically significant difference between treatment groups on the 0-10 verbal scale is 1.3.
Time Frame: 120 minutes
Measure: Mean (95% Confidence Interval); unit: units on a scale (0-10)
Arm/Group | IV Fluid Bolus | Control
Number analyzed (Participants) | 24 | 22
units on a scale (0-10) | 5.9 [4.8 to 7.1] | 5.5 [4.1 to 6.8]

3. Secondary Outcome: Percentage of Patients Free of Pain at 2 Hours
Description: Percentage of patients in each group who are pain-free two hours after initiation of the study intervention.
Time Frame: 120 minutes
Measure: Number; unit: percentage of participants
Arm/Group | IV Fluid Bolus | Control
Number analyzed (Participants) | 24 | 22
percentage of participants | 38 | 32

4. Secondary Outcome: Percentage of Patients With no or Mild Functional Disability Due to Headache at 60 Minutes
Description: Percentage of patients with functional disability due to headache rated as none or mild (able to perform all activities of daily living, but with some difficulty) at 60 minutes
Time Frame: 60 minutes
Measure: Number; unit: percentage of participants
Arm/Group | IV Fluid Bolus | Control
Number analyzed (Participants) | 25 | 24
percentage of participants | 72 | 75

5. Secondary Outcome: Percentage of Patients Who Would Want the Same IV Fluid Treatment on a Future Visit
Description: Percentage of participants answering "yes" to the question: "The next time you visit the ED with a headache, would you wish to receive the same IV fluid treatment again?"
Time Frame: 48 hours
Measure: Number; unit: percentage of participants
Arm/Group | IV Fluid Bolus | Control
Number analyzed (Participants) | 24 | 21
percentage of participants | 79 | 67

6. Secondary Outcome: Percentage of Patients Who Needed Rescue Medications
Description: Need for additional medications for pain control as determined by the treating physician.
Time Frame: 120 minutes
Measure: Number; unit: percentage of participants
Arm/Group | IV Fluid Bolus | Control
Number analyzed (Participants) | 24 | 22
percentage of participants | 21 | 32

7. Secondary Outcome: Length of Stay
Description: Length of emergency department stay
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | IV Fluid Bolus | Control
Number analyzed (Participants) | 25 | 24
minutes | 309 (68) | 316 (93)

8. Secondary Outcome: Verbal Pain Score at 48 Hours
Description: Current pain as reported by participants at 48 hour follow-up (0-10 verbal scale; 0 = No Pain, 10 = Maximum Pain).
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: units on a scale (0-10)
Arm/Group | IV Fluid Bolus | Control
Number analyzed (Participants) | 24 | 21
units on a scale (0-10) | 2.6 (3.3) | 1.9 (2.5)

9. Secondary Outcome: Percentage of Patients Reporting no Nausea or Mild Nausea at 60 Minutes
Description: Patients reporting no nausea or mild nausea
Time Frame: 60 mins
Measure: Number; unit: percentage of participants
Arm/Group | IV Fluid Bolus | Control
Number analyzed (Participants) | 25 | 24
percentage of participants | 88 | 96

10. Other Pre Specified Outcome: Verbal Report of Insertion Site Pain Score at 60 Minutes
Description: Pain at IV insertion site (0 = No Pain, 10 = Maximum Pain)
Time Frame: 60 minutes
Measure: Mean (Standard Deviation); unit: units on a scale (0-10)
Arm/Group | IV Fluid Bolus | Control
Number analyzed (Participants) | 24 | 22
units on a scale (0-10) | 0.42 (0.97) | 0.73 (1.32)

ADVERSE EVENTS:
Time Frame: 48 hours
Arm/Group | IV Fluid Bolus | Control
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24
Other Adverse Events (participants affected / at risk) | 0/25 | 0/24

LIMITATIONS AND CAVEATS:
This was a small-scale pilot study. The wide confidence intervals we observed do not exclude the possibility of a clinically relevant treatment effect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-08): https://cdn.clinicaltrials.gov/large-docs/60/NCT02933060/Prot_SAP_000.pdf